CLINICAL TRIAL: NCT03432182
Title: Characterization of Movements Occurring During Sleep in Very Premature Neonates: Relationship With Neurodevelopmental Outcome
Brief Title: Body Movements Analysis During Sleep in Very Premature Infants
Acronym: DODOPREMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A02687-46
Record Dates: First submitted 2018-02-01; First posted 2018-02-14 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Sleep
Keywords: Premature infant; sleep state; body movement; neurodevelopmental outcome
MeSH Terms: conditions — Premature Birth | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- very premature infants (Other): Electroencephalography allowing sleep observation
  Interventions: Diagnostic Test: electroencephalography

INTERVENTIONS:
Diagnostic Test: electroencephalography — Sleep states definition by electroencephalograpy

SUMMARY:
Sleep is a key factor for normal brain development of the newborn. However, it is poorly studied and little is known about its characterization, especially in premature infants. Body movements during sleep are easy to evaluate but studies on their relationship to normal sleep states are scarce and limited. This project aims to characterize body movements during sleep, assessed by electroencephalography, in very premature infants. Then, a correlation between body movements, sleep organization and neurodevelopmental outcome will be evaluated at 3 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 26 and 32 weeks gestation

Exclusion Criteria:

* Genetic abnormality
* Neurological pathology such as intraventricular hemorrhage > grade 2
* Any medication know for altering electroencephalography recording

Ages: 10 Days to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Body movements evaluation during sleep | 3 months
  number of movements observed according to sleep states

SECONDARY OUTCOMES:
Sleep states organization | 3 months
  sleep states characterization by electroencephalography according to postmenstrual age
Type of movements observed during sleep | 3 months
  Movements characterization according to sleep states
Neurodevelopmental outcome | 3 years
  neuropsychomotor evaluation by Bayley psychometric test

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Hospital CHRU, Nancy, France